CLINICAL TRIAL: NCT05164315
Title: Comparison of Oncologic Outcomes Between Tailored Surgery According to Intraoperative Local Excision Biopsy Versus Total Mesorectal Excision in ycT2-3N0M0 on Magnetic Resonance Imaging After Neoadjuvant Chemoradiotherapy for Low Rectal Cancer
Brief Title: Comparison Between Tailored Surgery Versus Total Mesorectal Excision in ycT2-3N0M0
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the high proportion of patients requiring TME(control group) suggests that proceeding with a randomized prospective clinical trial may not be feasible.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2107-697-002
Record Dates: First submitted 2021-11-29; First posted 2021-12-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer, Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored surgery (Experimental): Arm 1 will receive tailored surgery. If there are no cancer cells or the margin is negative in the local excision/biopsy during surgery, the operation will be terminated. And if the final pathology result is T2-4, or cancer cells and margin are positive in the frozen section during surgery, or the result of digital rectal examination and visual examination using anoretractor under general anesthesia is not suitable for local excision (visible and palpable tumor nodules), a total mesorectal excision will be performed.
  Interventions: Procedure: Tailored surgery
- Total mesorectal excision (TME) (Active Comparator): Arm 2 will receive TME. Surgery including high ligation of the inferior mesenteric artery and total mesorectal excision will be performed under the lithotomy position. After pelvic dissection, double-stapled anastomosis or transanal anastomosis will be performed, followed by diverting stoma. Abdominoperineal resection with permanent stoma is included.
  Interventions: Procedure: Total mesorectal excision (TME)

INTERVENTIONS:
Procedure: Tailored surgery — Procedure: Tailored surgery based on intraoperative local excision/biopsy
  Arms: Tailored surgery
Procedure: Total mesorectal excision (TME) — Procedure: Total mesorectal excision for all allocated patients
  Arms: Total mesorectal excision (TME)

SUMMARY:
The purpose of this study is to show that tailored treatment based on local excision can expand the target of non-radical treatment in ycT2-3N0M0 patients after neoadjuvant chemoradiotherapy for low rectal cancer and that the oncologic safety is not inferior to that of total mesorectal excision.

DETAILED DESCRIPTION:
Target number of subjects and calculation basis This study aims to show that the tailored treatment based on intraoperative local excision/biopsy is not oncologically inferior to total mesorectal excision. The 5-year overall survival rate expected from the existing standard treatment was 85% (van der Valk. 2018, Rullier. 2020). The non-inferior margin of the customized treatment was 10%, type 1 error 0.10, power 80%, 1:1 ratio. When calculated with a 10% dropout rate, a total of 346 people, 173 in each group, needs to be recruited.

Study Subject Recruitment Plan

1. Selection and enrollment of subjects: Subjects in clinical trials must be enrolled by the investigator before starting surgical treatment.
2. Document consent: To the patient who is considered to be able to participate in the clinical trial as a subject, an oral explanation of this clinical trial will be presented to the participants, and the written consent to participate in the clinical trial shall be obtained.
3. Preoperative evaluation A pre-treatment examination to determine the selection of subjects and their underlying condition will be conducted. Pre-treatment examination will be performed to review whether the subject meets the selection and exclusion criteria, and subjects with significant abnormalities will be excluded.

Control group setting and randomization method Tailored treatment based on local excision and total mesorectal excision are randomly assigned 1:1 by web-based random number table (REDCap).

Statistical Analysis The statistical analyses will be conducted using intention-to-treat, and per-protocol approaches. Multiple imputation for missing covariates will be performed to determine whether there are systematic differences in terms of missing data. Analyses of the primary and secondary outcomes will be adjusted for potential co-variates.

Results of the quality of life and sexual/urinary function questionnaires will be compared using linear generalized estimating equations (GEE), adjusted for baseline values, the time effect, and the interaction effect between time and treatment.

Clinical and pathological variables will be compared using χ2 tests or Fisher's exact test for categorical variables, or with Student's t-test for continuous variables. Disease-free survival, relapse-free survival, and overall survival curves will be plotted using the Kaplan-Meier method, and differences in survival curves will be compared using the log-rank test. Multivariable analyses using the Cox regression hazard model will be conducted to identify the factors that are independently associated with disease-free survival, relapse-free survival, and overall survival. All statistical tests will be two-sided and values of p<0·05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the rectum (AV≤5cm)
* Clinical ycT2-3N0 based on MRI after neoadjuvant chemoradiotherapy (including long/short-course chemoradiotherapy, total neoadjuvant therapy etc…)
* No evidence of distant metastases
* No prior pelvic radiation therapy
* No prior chemotherapy or surgery for rectal cancer
* Age 18 to 80 years
* No active infections requiring systemic antibiotic treatment (oral antibiotics are acceptable at the discretion of the treating physician)
* Women with childbearing potential who are negative for pregnancy test (urine or blood) and who agree to use effective contraceptive method. A woman of childbearing potential is defined of one who is biologically capable of becoming pregnant. Reliable contraception should be used from trial screening and must be continued throughout the study.
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study. Patients who do not read or understand Korean are eligible and may be consented according to institutional and federal regulations.
* Hemoglobin ≥ 10 g/dl (after correction for simple iron deficiency anemia), White blood cells ≥ 4,000/mm3, Platelets ≥ 100,000/mm3, Creatinine ≤ 1.5 mg/dl
* No significant dysfunction in the heart or lungs: When it is judged that the risk related to surgery due to functional impairment is not high during consultation treatment

Exclusion Criteria:

* Metastasis to the liver, lung, brain, bone, abdominal aortic lymph node, subclavian lymph node, inguinal lymph node, etc. at the time of evaluation before treatment
* Patients with a history of a prior malignancy
* Patients with serious heart disease and heart failure, severe lung disease or pulmonary insufficiency, active bacterial infection requiring parenteral antibiotic administration and/or other serious medical conditions
* Patients with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study.
* When it is legally impossible to participate in a clinical trial
* Patients who are pregnant or lactating
* When existing diseases and disorders are expected to affect the quality of life evaluation after surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years
  The percentage of people in a study or treatment group who are alive five years after their diagnosis or the date of randomization

SECONDARY OUTCOMES:
Immediate postoperative index | postoperative 30 days
  Postoperative recovery index, surgery-related complications, and mortality comparison (Clavien-Dindo classification III-V), histopathologic examination of the proximal/distal/peripheral margins
Oncologic outcomes | 5 years
  Rate of Disease-free Survival/Relapse-free Survival/Stoma-free Survival/Regrowth-free Survival through physical examination including digital rectal examination, carcinoembryonic antigen test (CEA), liver function test (AST/ALT), chest and abdominal CT and colonoscopy
Quality of Life evaluation | Conduct a survey before surgery and every year after surgery until the 3rd year
  The Korean version of EORTC QLQ 30 which is an evaluation instrument for the quality of life of cancer patients, and the Korean version of EORTC QLQ-CR29 which is an evaluation instrument for the quality of life of colon cancer patients.
Sexual/urination function evaluation | Conduct a survey before surgery and every year after surgery until the 3rd year
  IPSS (International Prostate Symptom Score) for urinary function test, IIEF-5 (5-item Version of the International Index of Erectile Function) for male sexual function test, FSFI (Female Sexual Function Index) for female sexual function test.
defecation function | Conduct before surgery and at 1, 2, and 3 years after surgery, (at 1, 2, and 3 years after stoma restoration).
  MSKCC questionnaire, fecal incontinence severity index (FISI), low anterior resection syndrome (LARS) score questionnaire and fecal incontinence quality of life index (FIQL), manometry

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea